CLINICAL TRIAL: NCT00037011
Title: Phase I Study of Oral Beta-Glucan and Intravenous Anti-GD2 Monoclonal Antibody 3F8 Among Patients With Metastatic Neuroblastoma
Brief Title: Beta-Glucan and Monoclonal Antibody in Treating Patients With Metastatic Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 01-075; P30CA008748 (NIH); MSKCC-01075; NCI-G02-2067
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — beta-Glucans; humanized 3F8 anti-GD2 monoclonal antibody

INTERVENTIONS:
Biological: beta-glucan
Biological: monoclonal antibody 3F8

SUMMARY:
RATIONALE: Biological therapies such as beta-glucan use different ways to stimulate the immune system and stop cancer cells from growing. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining beta-glucan and monoclonal antibody may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining beta-glucan and monoclonal antibody in treating patients who have metastatic neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of beta-glucan and monoclonal antibody 3F8 in patients with metastatic neuroblastoma.
* Determine the toxicity of this regimen in these patients.
* Assess the biological effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral beta-glucan and monoclonal antibody 3F8 (MOAB 3F8) IV within 1.5 hours on days 1-5 and 8-12. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of beta-glucan and MOAB 3F8 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

Patients are followed monthly for 6 months, every 2 months for 6 months, and then every 3-6 months for 2 years.

PROJECTED ACCRUAL: A maximum of 24 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-risk stage 4 metastatic neuroblastoma

  * May be confirmed by bone marrow involvement and elevated urinary catecholamines
* Progressive or persistent disease after intensive conventional chemotherapy that included induction with N6, N7, N8, or COG protocol with or without bone marrow or stem cell transplantation
* Poor long-term prognosis as defined by any of the following:

  * N-myc amplification in tumor cells
  * Diploid chromosomal content plus 1p loss of heterozygosity in tumor cells
  * Distant skeletal metastases
  * Unresectable primary tumor infiltrating across the midline
  * More than 10% tumor cells in bone marrow
* Measurable or evaluable disease documented at least 4 weeks after completion of prior systemic therapy

PATIENT CHARACTERISTICS:

Age:

* Under 50

Performance status:

* Not specified

Life expectancy:

* See Disease Characteristics

Hematopoietic:

* Platelet count greater than 25,000/mm^3
* Absolute neutrophil count greater than 500/mm^3

Hepatic:

* Not specified

Renal:

* Creatinine clearance greater than 60 mL/min

Other:

* No severe major organ toxicity
* No active life-threatening infections
* No prior allergy to mouse proteins
* No prior allergy to beta-glucan, oats, barley, mushrooms, or yeast
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior exposure to mouse antibodies and human anti-mouse antibody greater than 1,000 ELISA units/mL

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent supplemental beta-glucan either as food (e.g., bran cereals) or as complementary medicine

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2001-11; Primary Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Kong V. Cheung, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States